CLINICAL TRIAL: NCT00069186
Title: A Phase III, Multi-Center, Double-Blind, Placebo Controlled, Randomized Study of Creatine Monohydrate in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Study of Creatine Monohydrate in Patients With Amyotrophic Lateral Sclerosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Avicena Group (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AGI-ALS-III-01; Orphan Drug:01-1527
Record Dates: First submitted 2003-09-17; First posted 2003-09-23 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-04

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: Amyotrophic Lateral Sclerosis; ALS; Creatine; Creatine Monohydrate; Muscle Strength
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Creatine

INTERVENTIONS:
Drug: Creatine Monohydrate

SUMMARY:
The purpose of this study is to determine whether nine months of administration of creatine monohydrate results in an increase in muscle strength in patients with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
Introduction: Twenty-one ALS patients were enrolled in a placebo controlled pilot study at the Carolinas Neuromuscular/ALS-MDA Center, The University of Texas Health Science Center at San Antonio and The University of New Mexico at Albuquerque. At all time points sampled over a nine month period, patients taking creatine monohydrate had either a significantly greater improvement in their strength or a more modest decline compared to the patients taking placebo. Overall analysis of variance is significant for both an effect of the drug (p=0.002) and time (p< 0.001).The pilot study also showed that quality of life, as measured by ALSFRS-R, correlated significantly with the observed changes in muscle strength (MVIC).

Phase III Study: The primary objective of this study is to determine whether treatment with creatine monohydrate results in an increase in muscle strength relative to placebo in patients with amyotrophic lateral sclerosis (ALS), after three months, and at the end of a nine-month treatment period.

The study is a Phase III, eight-center, double-blind, placebo-controlled, randomized clinical trial designed to evaluate the safety and efficacy of creatine monohydrate in patients fulfilling the eligibility criteria. The subjects (n=156) will be randomized in a 1:1 ratio to receive treatment of highly purified creatine monohydrate or placebo (Dextrose, USP) for nine months. The subjects will be administered 10 grams of creatine monohydrate per day for the first five days, and then 5 grams per day thereafter. Each subject will be followed for the nine-month treatment period.

The primary outcome measure for the study is change in upper extremity motor function after three weeks, and at the end of a nine-month treatment period as tested by MVIC. Strength in ten arm muscles will be measured (bilateral shoulder and elbow flexion/extension and grip).

Patient safety will be assured by ongoing review of reports of adverse events, clinical laboratory data, and measurement of vital signs. These tests include: measurement of MVIC and muscle fatigue, measurement of FVC, completion of ALSFRS-R and SF-12 quality of life instruments, review of potential adverse effects, determination of vital signs and weight, serum creatinine and BUN, and urine dipstick for protein.

ELIGIBILITY:
* A clinical diagnosis of probable or definite lab-supported ALS, either SALS or FALS, according to modified El Escorial criteria.
* Males or females, 21 to 80 years of age.
* Patients receiving treatment with Rilutek® (riluzole) must be on a stable dose for at least 30 days immediately prior to enrollment.
* Women of childbearing potential must be non-lactating and surgically sterile or using an effective method of birth control (double barrier or oral contraception) and have a negative pregnancy test. Women will be considered menopausal if they have not had a menstrual cycle (period) for two years.
* Disease duration less than five years since symptom onset.
* At least 5 of 10 testable upper extremity muscle groups of MRC grade 4 or better.
* The patient must have given informed consent that has been approved by the appropriate Institutional Review Board (IRB).

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107
Dates: Start 2003-06; Study Completion 2005-04

PRIMARY OUTCOMES:
Change in upper extremity motor function after 3 weeks
Change in upper extremity motor function after 9 months

SECONDARY OUTCOMES:
Acute changes in muscle strength
Chronic changes in muscle strength
ALS functioning
Quality of life
Pulmonary function
Muscle fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Rosenfeld Jeffrey, MD, Principal Investigator — Carolinas ALS Center
Locations (8):
- United States (8):
  - University of California, San Francisco, San Francisco, California
  - University of Kansas, Kansas City, Kansas
  - University of New Mexico, Albuquerque, New Mexico
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Oregon Health Sciences University, Portland, Oregon
  - University of Texas Health Science Center, San Antonio, Texas
  - University of Virginia Health System, Charlottesville, Virginia